CLINICAL TRIAL: NCT02293343
Title: 24 Hrs Histamine Profile in Healthy Persons and Patients With Food Intolerance: Correlations Between Subjective Affliction and Measured Histamine Parameter
Brief Title: 24 Hrs Histamine Profile in Healthy Persons and Patients With Food Intolerance
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: Histamine profile 1
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Allergy; IBS
Keywords: histamine profile; IgE Antibodies
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- control group: healthy subjects
  Interventions: Other: blood profile
- IgE positive: patients with high IgE level in serum
  Interventions: Other: blood profile
- IBS patients: patients with afflictions, but no high IgE level and suspicion on histamine intolerance
  Interventions: Other: blood profile

INTERVENTIONS:
Other: blood profile

SUMMARY:
Over 24 hrs serum and plasma samples were collected every 3 hrs. With this a day histamine profile was created. 15 healthy persons with 20 patients with a high level of IgE in serum and 20 patients with afflictions but no high IgE level were compared. Measurment of histamine in plasma, urine and stool were realized. In addition to that Diaminoxidase, TNF alpha and IgE Antibodies were measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* appropriate invalid persons

Exclusion Criteria:

* pregnant and weaning persons

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects, patients with high IgE level and patients with afflictions, but no high IgE level
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Histamine | 24 hrs

SECONDARY OUTCOMES:
diaminoxidase | 24 hrs

OTHER OUTCOMES:
TNF alpha | 24 hrs
IgE | 24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Pinzer TC, Tietz E, Waldmann E, Schink M, Neurath MF, Zopf Y. Circadian profiling reveals higher histamine plasma levels and lower diamine oxidase serum activities in 24% of patients with suspected histamine intolerance compared to food allergy and controls. Allergy. 2018 Apr;73(4):949-957. doi: 10.1111/all.13361. Epub 2017 Dec 15. PMID 29154390